CLINICAL TRIAL: NCT00036465
Title: A Phase II, Randomized, Controlled, Pilot Study of Antiretroviral Switch at Lower Versus Higher HIV-1 RNA Levels in Subjects Experiencing Virologic Relapse on a Current HAART Regimen
Brief Title: Effects of Changing HIV Therapy at Lower Versus Higher Viral Loads
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: A5115; AACTG A5115; ACTG A5115; 10933 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2002-05-10; First posted 2002-05-13 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections
Keywords: Pilot Projects; HIV-1; RNA, Viral; Genotype; Viral Load; Antiretroviral Therapy, Highly Active; Treatment Experienced
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Behavioral: Treatment regimen change

SUMMARY:
This study will look at people who have been taking anti-HIV drugs but still have detectable levels of HIV. The purpose of the study is to find out what happens in those people who change anti-HIV drugs when their viral load reaches 200 copies compared to those who change anti-HIV drugs when their viral load reaches 10,000 copies. This study will also look at drug resistance (how well HIV responds to drugs), viral fitness (how well drug-resistant HIV copies itself), and immunologic reconstitution (how well the immune system recognizes various infections, including HIV).

Many patients experience virologic relapse (increase in viral load after sustained viral load suppression) within 1 to 2 years of taking anti-HIV drugs. The approach to treatment for patients who experience virologic relapse while on a highly active antiretroviral therapy (HAART) has not been defined. Current guidelines recommend switching to a new treatment regimen as soon as possible to prevent HIV from becoming even more resistant to anti-HIV drugs. However, there is evidence that patients can benefit from staying on the same HAART drugs, even after virologic relapse. This study wants to find what happens when drugs are changed immediately after virologic relapse (when the viral load is lower) compared to what happens if drugs are changed only after a delay (when the viral load is higher).

DETAILED DESCRIPTION:
Virologic relapse occurs within 1 to 2 years of antiretroviral therapy in up to 50 percent of HIV-infected individuals. The best treatment approach for patients who experience virologic rebound while on highly active antiretroviral therapy (HAART) has not been defined. Current guidelines recommend switching to a new treatment regimen shortly after virologic rebound in an effort to avoid sequential accumulation of multiple resistance mutations. However, early treatment switching has numerous disadvantages: risk of virologic rebound on the new therapy, a limited number of drug combinations available to treat such rebounds, and difficulty in obtaining early genotypic and phenotypic drug-resistance information to guide treatment modification. Delaying a switch to a new antiretroviral regimen has the advantage of preserving future treatment options, and HIV levels may remain partially suppressed even after drug-resistant mutants emerge. Moreover, several observational studies describe maintenance of immunologic and clinical benefits of HAART even after virologic rebound. Delayed treatment switches, however, raise concerns about sequential accumulation of drug resistance mutations that may diminish the chances of viral resuppression with successive HAART regimens, and the long-term immune consequences of virologic rebound on HAART are not known. It is therefore important to evaluate the viral and immunologic responses among patients randomized to either an early or delayed HAART switch.

This study enrolls patients who have a viral load of at least 200, but less than 10,000 copies/ml. The patients are randomized into 2 treatment arms. Arm A (immediate switch) patients have genotypic resistance testing at entry. Based on the resistance test results, their antiretroviral treatment regimen is modified to a switch treatment regimen. Switch treatment initiates no later than Week 4. Arm B (delayed switch) patients continue their current antiretroviral regimen and have genotypic resistance testing when their plasma HIV-1 RNA levels reach 10,000 copies/ml or greater. Based on the resistance test results, their antiretroviral treatment regimen is modified to a switch treatment regimen. Switch treatment initiates no later than 4 weeks from the date of at least 10,000 copies/ml viral load, or from the date of an absolute CD4 count reduced by 20 percent from baseline value. Patients who never meet the switch criteria remain on study.

All patients are followed for a minimum of 48 weeks after entry. No antiretroviral drugs are provided by the study.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-infected.
* Have a CD4 cell count of 200 cells/mm3 or more within 45 days prior to entry.
* Are currently receiving the same HAART regimen for at least 4 months.
* Had a documented viral load of less than 500 copies/ml at any time prior to screening on the current stable antiretroviral regimen.
* Have a detectable plasma viral load on current stable anti-HIV regimen, as defined in the protocol, within 52 weeks prior to screening.
* Are willing to remain on their current regimen until their scheduled switch.
* Have a negative pregnancy test within 48 hours prior to entry.
* Are at least 13 years old.
* Agree not to participate in the conception process (active attempts to become pregnant or to make someone pregnant) while on study and for 60 days after going off study.
* Agree to use 2 acceptable forms of contraception while on study and for 60 days after going off study.

Exclusion Criteria

Patients may not be eligible for this study if they:

* Do not adhere with current antiretroviral therapy.
* Have an infection or cancer that requires treatment within 45 days prior to entry.
* Are pregnant or breast-feeding.
* Have used any experimental agents, systemic corticosteroids, or drugs that interfere with the immune system within 45 days prior to entry.
* Have received any HIV vaccine within 90 days prior to entry.
* Use drugs or alcohol that, in the opinion of the investigator, would interfere with the study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Riddler, Study Chair
Locations (23):
- United States (23):
  - Willow Clinic, Menlo Park, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor General/UCLA, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Harvard (Masschusetts General Hosp), Boston, Massachusetts
  - Brigham and Womens Hosp, Boston, Massachusetts
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown Univ / Miriam Hosp, Providence, Rhode Island
  - Miriam Hosp / Brown Univ, Providence, Rhode Island
  - Comprehensive Care Clinic / Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Texas, Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Derived] Riddler SA, Jiang H, Tenorio A, Huang H, Kuritzkes DR, Acosta EP, Landay A, Bastow B, Haas DW, Tashima KT, Jain MK, Deeks SG, Bartlett JA. A randomized study of antiviral medication switch at lower- versus higher-switch thresholds: AIDS Clinical Trials Group Study A5115. Antivir Ther. 2007;12(4):531-41. doi: 10.1177/135965350701200415. PMID 17668562